CLINICAL TRIAL: NCT00227084
Title: Effect of Arista AH-Haemostatic Powder in Plastic Surgery. A Prospective, Consecutive Randomized Study in 30 Women Undergoing Reduction of Both Mamma
Brief Title: Effect of Arista Powder on Bleeding in Reductive Mammary Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Ullevaal University Hospital (Other); Medafor (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1.2005.419
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Mammaplasty
Keywords: Mammary glands; hemostasis; Mammaplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Arista AH hemostasis powder

SUMMARY:
To evaluate whether Arista AH which contains microporous polysaccharides used as a powder applied to the wound area during mammary surgery reduces the amount of bleeding and the duration of surgery. Both mammae are operated on in the same procedure, and one side without Arista serves as control side

DETAILED DESCRIPTION:
During the operation,before the first incision a randomization envelope is opened. Always starts on the same side, with or without Arista according to the envelope. After surgery, vacuum drains are placed and the amount of drained material and hgb content is measured 24 hours later by nursing staff blinded to what side had Arista.Patients scores postoperative pain with VAS score bilaterally.

Three months postoperatively the patients are checked by a physician blinded for what side had Arista

ELIGIBILITY:
Inclusion Criteria:

* All women for mammary hypertrophy day surgery. No exclusions in this group.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
duration of surgery
amount of bleeding on drain

CONTACTS AND LOCATIONS:
Overall Officials: Christian Askenberg, MD, Principal Investigator — Ullevaal University Hospital; Petter A Steen, MD,PhD, Study Director — University of Oslo
Locations (1):
- Ulleval University Hospital, Oslo, Norway